CLINICAL TRIAL: NCT04431739
Title: Differentiation Between Malignant and Benign Vertebral Bone Marrow Lesions by Diffusion Weighted Imaging (DWI) and Apparnt Diffusion Coefficient (ADC) Values
Brief Title: Vertebral Bone Marrow Lesions by DWI and ADC Values
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mohamed Ibrahim Abbas (Other)
Responsible Party: Sponsor-Investigator, Mohamed Ibrahim Abbas, MD, Assiut University
Organization: Assiut University (Other)
Other Study IDs: vertebral bone marrow lesions
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Vertebral Lesion
MeSH Terms: interventions — Diffusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI including conventional MRI, DWI with multiple ADC values — The utility of apparent diffusion coefficient obtained in diffusion-weighted MR imaging for the differentiation between benign and malignant vertebral lesions

SUMMARY:
The aim of the work is to assess the utility of apparent diffusion coefficient obtained in diffusion-weighted MR imaging for the differentiation between benign and malignant vertebral lesions.

DETAILED DESCRIPTION:
MRI has a high sensitivity in delineating the pathology, its specificity is low. Osteoporotic and metastatic compression fractures may be mistaken for each other in the acute phase (Wong and Suresh, 2018). Edema in the acute phase of benign fractures may replace normal bone marrow and cause hypointense signal changes in T1-weighted images and hyperintense signal changes in T2-weighted images, at the same time taking contrast material. These changes are also typical for metastasis and cause confusion in diagnosis when only one lesion is present (Mauch et al., 2018).

Diffusion-weighted imaging (DWI) has recently appeared as a new method of screening in characterizing lesions without necessitating contrast material and in evaluating the vertebrae quantitatively (Lee et al., 2019) Diffusion-weighted-imaging (DWI) provides microscopic information from water protons which is not possible using conventional magnetic resonance imaging (MRI) (Partridge et al., 2017). DWI measures the random (Brownian) extra, intra and transcellular motion of water molecules (Ahlawat and Fayad, 2018) Apparent-diffusion-coefficient (ADC) is a quantitative parameter calculated from DWI that combines the effects of capillary perfusion and water diffusion (Wang et al., 2018) In a comparatively small number of surveys, ADC values have been studied in discriminating the infectious lesions from the malign lesions The utility of apparent diffusion coefficient obtained in diffusion-weighted MR imaging for the differentiation between benign and malignant vertebral lesions, and to determine the sensitivity and the specificity in differentiating benign and malignant vertebral lesions according to the optimal cutoff ADC value (Dahnert et al., 2017)

ELIGIBILITY:
Inclusion Criteria:

After taking clinical complaint and Orthopedic and neurological examinations, all patients (any age or sex) with suspected bone marrow focal lesions will undergo DWI and ADC map.

Exclusion Criteria:

All patients who contraindicated for MRI study as patients with cardiac pacemaker, any metallic stent, claustrophobia and morbid obesity.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be subjected to the following:
  1. Clinical picture
  2. Orthopedic and neurological examination Imaging studies
     * MRI of spine (site of complain) (T1WIs and T2WIs).
     * Diffusion-Weighted Imaging (DWI) and apparent diffusion coefficient (ADC) mapping.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
The utility of apparent diffusion coefficient obtained in diffusion-weighted MR imaging | 6 months
  The utility of apparent diffusion coefficient obtained in diffusion-weighted MR imaging for the differentiation between benign and malignant vertebral lesions

SECONDARY OUTCOMES:
Sensitivity, specificity and predictive value of the procedure | 6 months
  Compared the results with histo-pathological biopsy and follow up studies after medical treatment to detect (sensitivity, specificity and predictive value) of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Abdel Kareem H Abdalla, MD, Study Chair — Professor of Radio-diagnosis, Faculty of Medicine -Assuit University

REFERENCES:
- [Result] Li K, Huang L, Lang Z, Ni L, Du J, Yang H. Reliability and Validity of Different MRI Sequences in Improving the Accuracy of Differential Diagnosis of Benign and Malignant Vertebral Fractures: A Meta-Analysis. AJR Am J Roentgenol. 2019 Aug;213(2):427-436. doi: 10.2214/AJR.18.20560. Epub 2019 Apr 30. PMID 31039028
- [Result] Mauch JT, Carr CM, Cloft H, Diehn FE. Review of the Imaging Features of Benign Osteoporotic and Malignant Vertebral Compression Fractures. AJNR Am J Neuroradiol. 2018 Sep;39(9):1584-1592. doi: 10.3174/ajnr.A5528. Epub 2018 Jan 18. PMID 29348133
- [Result] Lee K, Park HY, Kim KW, Lee AJ, Yoon MA, Chae EJ, Lee JH, Chung HW. Advances in whole body MRI for musculoskeletal imaging: Diffusion-weighted imaging. J Clin Orthop Trauma. 2019 Jul-Aug;10(4):680-686. doi: 10.1016/j.jcot.2019.05.018. Epub 2019 May 29. PMID 31316239